CLINICAL TRIAL: NCT01677520
Title: Investigation of Adipose-Derived Stem Cells in Human Lipoaspirate
Brief Title: Investigation of Stem Cells in Human Lipoaspirate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, William A. Zamboni, M.D., Professor and Chair Department of Surgery UNSOM, University of Nevada, Las Vegas
Other Study IDs: 12.08.004
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: adipose-derived stem cells; viable ADSCs; apoptosis; necrosis; cryopreservation
MeSH Terms: conditions — Breast Neoplasms; Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cells from lipoaspirate maximum of 20 days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 18-30 yrs, 31-50 yrs, 51-70 yrs: No intervention

SUMMARY:
The overall purpose of this study is to enhance identification and isolation of ADSCs and adipocytes, to find the optimum culturing conditions to increase growth and volume of grafts, and to study the effects of cryopreservation on ADSCs and adipocytes. Fat injections are used in aesthetic surgery but tend to disassemble over time. If the investigators can enhance growth and volume of fat in culture, the investigators could use fat grafts in reconstruction of cancer and traumatic injury defects with the patients own cultured fat cells and grafts.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18-70 yrs) who have scheduled surgical lipectomy of the hips, abdomen, or thighs are prospective subjects for this study.

Exclusion Criteria:

* Pregnant women will be excluded to protect the unborn child.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2011-03; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Percent of Viable ADSCs | Day of Surgery
  Percent of viable ADSCs will be measured on fresh samples and samples refrigerated for different times.

SECONDARY OUTCOMES:
Percent of Apoptotic ADSCs | Day of Surgery
  Percent of apoptotic ADSCs will be measured on fresh samples and on refrigerated samples at 1, 2, 3, and 4 days refrigerated storage.

OTHER OUTCOMES:
Percent of Necrotic ADSCs | Day of Surgery
  Percent of necrotic ADSCs will be measured on fresh samples and on refrigerated samples at 1, 2, 3, and 4 days of refrigerated storage.

CONTACTS AND LOCATIONS:
Overall Officials: William A Zamboni, M.D., Principal Investigator — UNSOM; Wei Z Wang, M.D., Study Director — wwang@medicine.nevada.edu
Locations (1):
- University of Nevada School of Medicine Patient Care Center, Las Vegas, Nevada, United States